CLINICAL TRIAL: NCT02240030
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Investigating the Efficacy and Safety of CVT 301 (Levodopa Inhalation Powder) in Parkinson's Disease Patients With Motor Response Fluctuations (OFF Phenomena) (SPAN-PD™)
Brief Title: Efficacy and Safety Study of CVT-301 In Parkinson's Disease Patients With OFF Episodes
Acronym: SPAN-PD™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-301-004
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Motor fluctuations; levodopa; inhaled drugs; OFF episodes
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CVT-301 Low Dose (Experimental): Capsules of levodopa inhalational powder used up to 5 times/day for OFF episodes for 3 months duration
  Interventions: Drug: CVT-301 Low Dose
- CVT-301 High Dose (Experimental): Capsules of levodopa inhalational powder used up to 5 times/day for OFF episodes for 3 months duration
  Interventions: Drug: CVT-301 High Dose
- Placebo (Placebo Comparator): Capsules of inhalation-grade lactose used up to 5 times/day for OFF episodes for 3 months duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CVT-301 Low Dose
  Other Names: Inhaled levodopa
  Arms: CVT-301 Low Dose
Drug: CVT-301 High Dose
  Other Names: Inhaled levodopa
  Arms: CVT-301 High Dose
Other: Placebo
  Other Names: Inhalation-grade lactose
  Arms: Placebo

SUMMARY:
This randomized, multicenter, placebo-controlled, double-blind study will evaluate the efficacy and safety of inhaled CVT 301 compared with placebo in PD patients experiencing motor response fluctuations (OFF phenomena) as an outpatient (i.e., at home) and in the clinic.

Patients who successfully complete this study will be eligible to enroll into a 12 month treatment extension (CVT-301-004E) study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (PD) diagnosed between the ages of 30 and 85 years;
* Hoehn and Yahr Stage 1-3 in an "on" state;
* Require levodopa-containing medication regimen at least 3 times during the waking day;
* Experience motor fluctuations with a minimum of 2 hours of average daily "off" time per waking day (excluding early morning "off" time) and demonstrate levodopa responsiveness;
* Are on stable PD medication regimen;
* Total daily LD dose <1600 mg/day;
* Able to perform a spirometry maneuver in the ON and OFF states;
* Normal cognition confirmed by MMSE score ≥25

Exclusion Criteria:

* Pregnant or lactating females;
* Previous surgery for PD or plan to have stereotactic surgery during the study period;
* History of psychotic symptoms requiring treatment, or suicide ideation or attempt within last year;
* Known contraindication to the use of levodopa;
* Any significant condition, severe concurrent disease, abnormality or finding that would make patients unsuitable or may compromise patient safety;
* Any contraindication to performing routine spirometry.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Oh, MD, Study Director — Acorda Therapeutics
Locations (74):
- United States (55):
  - Acorda Site #5020, Scottsdale, Arizona
  - Acorda Site #5042, Fresno, California
  - Acorda Site #5064, Fullerton, California
  - Acorda Site #5035, Loma Linda, California
  - Acorda Site #5027, Long Beach, California
  - Acorda Site #5037, Los Angeles, California
  - Acorda Site #5070, Pasadena, California
  - Acorda Site #5047, Reseda, California
  - Acorda Site #5068, Santa Ana, California
  - Acorda Site #5069, Torrance, California
  - Acorda Site #5052, Washington D.C., District of Columbia
  - Acorda Site #5046, Atlantis, Florida
  - Acorda Site #5053, Aventura, Florida
  - Acorda Site #5013, Boca Raton, Florida
  - Acorda Site #5016, Jacksonville, Florida
  - Acorda Site #5071, Maitland, Florida
  - Acorda Site #5044, Orlando, Florida
  - Acorda Site #5060, Palm Beach Gardens, Florida
  - Acorda Site #5001, Port Charlotte, Florida
  - Acorda Site #5065, St. Petersburg, Florida
  - Acorda Site #5012, Tampa, Florida
  - Acorda Site #5040, Atlanta, Georgia
  - Acorda Site #5025, Chicago, Illinois
  - Acorda Site #5030, Chicago, Illinois
  - Acorda Site #5011, Elk Grove Village, Illinois
  - Acorda Site #5003, Kansas City, Kansas
  - Acorda Site #5067, Baton Rouge, Louisiana
  - Acorda Site #5057, Baltimore, Maryland
  - Acorda Site #5056, Boston, Massachusetts
  - Acorda Site #5018, Boston, Massachusetts
  - Acorda Site #5002, Bingham Farms, Michigan
  - Acorda Site #5014, West Bloomfield, Michigan
  - Acorda Site #5041, Golden Valley, Minnesota
  - Acorda Site #5006, St Louis, Missouri
  - Acorda Site #5023, Las Vegas, Nevada
  - Acorda Site #5028, Albany, New York
  - Acorda Site #5039, Brooklyn, New York
  - Acorda Site #5031, New York, New York
  - Acorda Site #5032, New York, New York
  - Acorda Site #5004, New York, New York
  - Acorda Site #5038, Syracuse, New York
  - Acorda Site #5048, Charlotte, North Carolina
  - Acorda Site #5005, Cleveland, Ohio
  - Acorda Site #5050, Norwood, Ohio
  - Acorda Site #5062, Portland, Oregon
  - Acorda Site #5036, Allentown, Pennsylvania
  - Acorda Site #5010, Philadelphia, Pennsylvania
  - Acorda Site #5058, Willow Grove, Pennsylvania
  - Acorda Site #5022, Charleston, South Carolina
  - Acorda Site #5029, Nashville, Tennessee
  - Acorda Site #5019, Houston, Texas
  - Acorda Site #5045, Houston, Texas
  - Acorda Site #5049, Henrico, Virginia
  - Acorda Site #5059, Virginia Beach, Virginia
  - Acorda Site #5051, Kirkland, Washington
- Canada (3):
  - Acorda Site #5103, London, Ontario
  - Acorda Site #5104, Ottawa, Ontario
  - Acorda Site #5105, Toronto, Ontario
- Czechia (2):
  - Acorda Site #5201, Prague
  - Acorda Site #5203, Prague
- Poland (8):
  - Acorda Site #5304, Katowice
  - Acorda Site #5306, Krakow
  - Acorda Site #5303, Krakow
  - Acorda Site #5307, Krakow
  - Acorda Site #5302, Lodz
  - Acorda Site #5308, Warsaw
  - Acorda Site #5301, Warsaw
  - Acorda Site #5305, Zaspa
- Spain (6):
  - Acorda Site #5407, Pamplona, Navarre
  - Acorda Site #5404, Barcelona
  - Acorda Site #5406, Barcelona
  - Acorda Site #5405, Madrid
  - Acorda Site #5403, San Sebastián
  - Acorda Site #5401, Sant Cugat del Vallès

REFERENCES:
- [Derived] LeWitt PA, Hauser RA, Pahwa R, Isaacson SH, Fernandez HH, Lew M, Saint-Hilaire M, Pourcher E, Lopez-Manzanares L, Waters C, Rudzinska M, Sedkov A, Batycky R, Oh C; SPAN-PD Study Investigators. Safety and efficacy of CVT-301 (levodopa inhalation powder) on motor function during off periods in patients with Parkinson's disease: a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Neurol. 2019 Feb;18(2):145-154. doi: 10.1016/S1474-4422(18)30405-8. PMID 30663606
- See also: Click here for more information about this study: CVT-301-004 — http://cvt301.acordatrials.com/en/patient/?src=clinicaltrialsgov004

RESULTS

PARTICIPANT FLOW:
Groups:
- CVT-301 Low Dose; CVT-301 High Dose: Capsules of levodopa inhalational powder used up to 5 times/day for OFF episodes for 3 months duration
  CVT-301
- Placebo: Capsules of inhalation-grade lactose used up to 5 times/day for OFF episodes for 3 months duration.
  CVT-301
Period: Overall Study
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
Started | 113 | 114 | 112
Completed | 96 | 97 | 97
Not Completed | 17 | 17 | 15

BASELINE CHARACTERISTICS:
Population: 12 participants were randomized but withdrew before receiving any study drug (4 placebo, 2 CVT-301 low-dose, 6 CVT-301 high-dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo | Total
Number analyzed (Participants) | 113 | 114 | 112 | 339
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 58 | 55 | 167
  >=65 years | 59 | 56 | 57 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.24) | 63.5 (7.97) | 62.6 (8.83) | 63.3 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 26 | 90
  Male | 80 | 83 | 86 | 249
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9 | 2 | 9 | 20
  United States | 86 | 81 | 81 | 248
  Poland | 18 | 29 | 19 | 66
  Spain | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part III
Description: Primary Efficacy Analysis: Change from Predose in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score at 30 Minutes post-dose at Week 12 for CVT-301 High Dose versus Placebo (ITT Population). UPDRS Part III ranges from 0 minimum to 86 maximum, with lower scores indicating better movement. Units on a scale.
Time Frame: 30 minutes post-dose at week 12
Population: 12 participants were randomized but withdrew before receiving any study drug (4 placebo, 2 CVT-301 low-dose, 6 CVT-301 high-dose).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CVT-301 High Dose | Placebo
Number analyzed (Participants) | 114 | 112
units on a scale | -9.83 (1.506) | -5.91 (1.500)

2. Secondary Outcome: Proportion of Patients Achieving Resolution of an OFF to an ON State Within 60 Minutes.
Description: Examiner-assessed observation - Subject Achieving Resolution of an OFF to and ON state within 60 Minutes at TV4 - Observed
Time Frame: at week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
Number analyzed (Participants) | 113 | 114 | 112
Participants | 55 | 56 | 35

3. Secondary Outcome: UPDRS Part III Motor Score at 20 Minutes
Description: Change from Predose in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score at 20 Minutes post-dose at Week 12 for CVT-301 High Dose versus Placebo (ITT Population) and CVT 301 Low Dose versus Placebo. UPDRS Part III ranges from 0 minimum to 86 maximum, with lower scores indicating better movement. Units on a scale.
Time Frame: at week 12
Population: as for outcome 1
Measure: Least Squares Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
Number analyzed (Participants) | 113 | 114 | 112
units on a scale | -8.47 [-11.11 to -5.82] | -9.04 [-11.70 to -6.37] | -6.49 [-9.15 to -3.83]

4. Secondary Outcome: Proportion of Subjects Who Improved PGIC With CVT-301 vs. Placebo at Week 12
Description: Patient Global impression of change at treatment visit 4 (week 12) by improvement category. Seven point Likert scale ranging from 1= much worse to 7= much better.
Time Frame: week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
Number analyzed (Participants) | 113 | 114 | 112
Participants | 61 | 70 | 45

5. Secondary Outcome: UPDRS Part III at 10 Min.
Description: Change from Predose in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score at 10 Minutes post-dose at Week 12 for CVT-301 High Dose versus Placebo (ITT Population). UPDRS Part III ranges from 0 minimum to 86 maximum, with lower scores indicating better movement. Units on a scale.
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
Number analyzed (Participants) | 113 | 114 | 112
units on a scale | -5.16 [-7.31 to -3.00] | -6.45 [-8.62 to -4.27] | -4.18 [-6.35 to -2.01]

6. Secondary Outcome: PD Patient Diary
Description: Change in total daily OFF times for 3 consecutive days prior to week 12 visit compared to 3 consecutive days prior to baseline visit. Participants recorded On or Off state in 30 minute intervals during waking hours.
Time Frame: post week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
Number analyzed (Participants) | 113 | 114 | 112
hours | -0.58 [-1.13 to -0.03] | -0.47 [-1.02 to 0.09] | -0.48 [-1.03 to 0.08]

ADVERSE EVENTS:
Time Frame: 12 Week Study
Arm/Group | CVT-301 Low Dose | CVT-301 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/114 | 0/112
Serious Adverse Events (participants affected / at risk) | 6/113 | 2/114 | 3/112
Other Adverse Events (participants affected / at risk) | 37/113 | 44/114 | 10/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVT-301 Low Dose (N=113) | CVT-301 High Dose (N=114) | Placebo (N=112)
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Lumbar spinal stinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVT-301 Low Dose (N=113) | CVT-301 High Dose (N=114) | Placebo (N=112)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 17 | 2
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Upper respiratory tract (Infections and infestations) | 2 | 7 | 3
Dyskinesia (Nervous system disorders) | 5 | 4 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 5
Nausea (Gastrointestinal disorders) | 0 | 6 | 3
Fall (Injury, poisoning and procedural complications) | 5 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.